CLINICAL TRIAL: NCT01407562
Title: Phase I Study of Pazopanib in Combination With Weekly Paclitaxel and Carboplatin to Assess the Safety and Tolerability in Patients With Advanced Solid Tumors
Brief Title: Study of Pazopanib, Paclitaxel, and Carboplatin in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Nancy Chan, MD, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro0220110062; P30CA072720 (NIH); NCI-2011-02448 (Other: CTRP (Clinical Trails Reporting Program)); 051101 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2011-07-20; First posted 2011-08-02 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Unspecified Adult Solid Tumor - Protocol Specific; Breast Cancer - Female
MeSH Terms: interventions — pazopanib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib with paclitaxel and carboplatin (Experimental)
  Interventions: Drug: Pazopanib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pazopanib — Starting dose is 400 given on Days 2-5, 9-12, and 16-26 of each 28 day cycle
Drug: Paclitaxel — Starting dose is 60 mg/m2 IV on days 1, 8, and 15 of each 28 day cycle
Drug: Carboplatin — Starting dose of carboplatin that corresponds to an AUC of 2, IV on days 1, 8, and 15 of each 28 day cycle

SUMMARY:
This is an open label, dose escalation study to determine the safety and tolerability and maximum tolerated dose of pazopanib combined with weekly paclitaxel and carboplatin in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open label, dose escalation study to determine the maximum tolerated dose (MTD) of pazopanib combined with weekly paclitaxel and carboplatin in patients with advanced solid tumors. There will be a dose expansion cohort of thirty patients to assess detailed pharmacokinetics and to assess any signal of activity in patients with solid tumors and in a portion who have breast cancer that is triple negative (ER-negative, PR-negative, and HER2-negative).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a solid malignancy with advanced disease that has relapsed, that is refractory to standard therapies, or for which there is not standard therapy, or for which the patient opts not to receive standard therapy.
* At the recommended phase II dose level, triple-negative breast cancer defined as ER-negative, PR-negative, and HER2-negative, will be enrolled and another 10 patients with a solid malignancy who would benefit from a paclitaxel and carboplatin-based regimen, will also be enrolled.
* Male or female ≥ 18 years of age
* Able to swallow and retain oral medications

Exclusion Criteria:

* Major surgery within last 28 days or cytotoxic chemotherapy, biologic therapy, investigational agents, or radiotherapy within last 21 days. Patients who have completed therapy with mitomycin C or nitrosurea will have to wait 42 days.
* More than 3 prior lines of cytotoxic chemotherapy for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09-17 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of pazopanib with weekly paclitaxel and carboplatin on a 28- day cycle | 4 years, 6 months
  Toxicity will be assessed every 28 days up to 30 days after the last dose of treatment. Dose limiting toxicity is defined as
  1. Non-hematological toxicity ≥ grade 3 (excluding alopecia, nausea, vomiting, or diarrhea for which adequate supportive therapy has not been instituted).
  2. Hematologic toxicity:
     * Grade 4 neutropenia lasting ≥ 7 days
     * Grade 4 neutropenia and fever of ≥ 38.5°C
     * ≥ Grade 3 neutropenia with ≥ Grade 3 infection
     * Grade 4 thrombocytopenia
     * Inability to start next cycle of treatment by more than 4 weeks due to unresolved toxicity

SECONDARY OUTCOMES:
Determine the drug-drug interactions with paclitaxel, carboplatin, and pazopanib | 4 years, 3 months
  The first 15 patients enrolled in the dose expansion cohort will undergo PK sampling as this is felt to be an adequate sample size.
  4 blood samples (2 mL each) for the analysis of paclitaxel will be obtained in Cycle 1 Day 1 and Cycle 2 Day 1
  2 blood samples (2 mL each) for the analysis of carboplatin will be obtained in Cycle 1 Day 1 and Cycle 2 Day 1
  1 blood sample (2 mL) for the analysis of pazopanib will be collected in Cycle 2 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chan, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No